CLINICAL TRIAL: NCT07156032
Title: Evaluation of the Effect of Computer Controlled Starpen Automatic Injection Device Versus Conventional Syringe on Pain Perception During Infiltration Anesthesia and Extraction of Maxillary Primary Molars : A Randomized Clinical Trial
Brief Title: Effect of Starpen Injection Device Versus Conventional Syringe During Anesthesia and Extraction of Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghadeer Mohamed Sayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPen device injection in MPM
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Pain Perception of the New Device
Keywords: Starpen device; Computer controlled automatic injection device; Computer controlled injection; pain perception; infiltration anesthesia; extraction of maxillary primary molars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Starpen automatic injection device (Experimental): effect of computer controlled Starpen device on pain perception during infiltration anesthesia and extraction of maxillary primary molars
  Interventions: Device: Starpen automatic injection device
- Conventional syringe (Active Comparator): Conventional syringe on pain perception during infiltration anesthesia and extraction of maxillary primary molars
  Interventions: Procedure: conventional syringe

INTERVENTIONS:
Device: Starpen automatic injection device — Starpen device will be used on high speed 45-150s with the conventional carpule of articaine HCL 4% with 1:100,000 epinephrine and short needle
  Other Names: computer controlled injection device
  Arms: Starpen automatic injection device
Procedure: conventional syringe — injection will be done using conventional metal syringe with articaine HCL 4% with 1:100,000 epinephrine and short needle
  Other Names: dental syringe
  Arms: Conventional syringe

SUMMARY:
To evaluate the effect of Starpen device on pain perception during anesthesia and extraction of maxillary primary molars.

DETAILED DESCRIPTION:
After enrollment of the patients according to the eligibility criteria, taking full medical , dental history and informed consents from the parents. Clinical and radiographic examination will be done for the tooth to be extracted. A diagnostic chart with personal, medical and dental history will be filled out . Also preoperative psychological management of the child through positive reinforcement techniques should be done . Then the two parallel groups will have local anesthesia using an infiltration technique in the upper jaw ; one group with conventional syringe and the other group by Starpen automatic injection device . Both groups will have the site of injection well prepared before injection by the same way and technique. In Addition, procedures as anesthesia injection and extraction will be done according to the guidelines set by the American Academy of Pediatric Dentistry . After the procedure is done , the participants and their parents will be instructed about post-operative care and the need of a space maintainer will be taken into account. Moreover subjective and objective pain will be assessed and scored during procedure of anesthesia injection and extraction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-8 years
* Cooperative children ( rating 3 or 4 based on the Frankl behavior scale )
* Medically fit children (ASA I )
* Children mentally capable of communication
* First dental visit
* Patient requiring extraction of upper primary molars due to root caries , crown fractures, periapical disease and failed pulpotomies
* No acute dental pain

Exclusion Criteria:

* Children with a behavioral management problem
* Parental refusal of participation
* Children with previous history of local anesthesia injection
* Medically unfit children (other than ASA I )
* Uncooperative children ( other than Frankl 3,4)
* Children under medications ( antibiotics and analgesics ) for the previous 48 hours that could alter the pain perception
* Teeth that showed any signs of mobility , ankylosis or root resorption affecting more than one third the root
* Acute dental pain

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Subjective pain during injection | during procedure
  Subjective pain perception during injection of infiltration anesthesia using Wong Baker Scale which represents a series of faces from 0-value happy face that represents lack of pain to a 10-value crying face which represents the worst possible face . On this basis , the patient chooses the face that best describes his/her level of pain.

SECONDARY OUTCOMES:
Objective pain during infiltration | during procedure
  Objective pain perception during infiltration anesthesia using Faces, legs, Arms, Crying, Consolability (FLACC) scale . The scale is scored in a range of 0-10 with 0 representing no pain. The observation lasts for 2-5 minutes. Each parameter is evaluated on a scale from 0 to 2; the total score is interpreted as follows: 0 = relaxed and comfortable, 1-3=mild, 4-6=moderate pain, 7-10=severe discomfort/ pain.
Subjective pain during extraction | during procedure
  Subjective pain perception during extraction of maxillary primary molars using Wong Baker Scale which represents a series of faces from 0-value happy face that represents lack of pain to a 10-value crying face which represents the worst possible face . On this basis , the patient chooses the face that best describes his/her level of pain.
Objective pain during extraction | during procedure
  Objective pain perception during extraction of maxillary primary molars using Faces, legs, Arms, Crying, Consolability (FLACC) scale . The scale is scored in a range of 0-10 with 0 representing no pain. The observation lasts for 2-5 minutes. Each parameter is evaluated on a scale from 0 to 2; the total score is interpreted as follows: 0 = relaxed and comfortable, 1-3=mild, 4-6=moderate pain, 7-10=severe discomfort/ pain.
Physiological parameters ( heart rate ) | Readings will be taken before and during anesthesia injection and during extraction.
  Physiological parameters ( heart rate) at three time points : baseline , during injection and during extraction using pulse oximeter on the child's index finger. At which 70-100 bpm is the normal range at rest and higher heart rate readings reflects anxiety/pain/ discomfort .
Physiological parameter ( oxygen saturation) | Readings will be taken before and during anesthesia injection and during extraction.
  Physiological parameter ( oxygen saturation) at three time points : baseline , during injection and during extraction using pulse oximeter on the child's index finger. At which 95-100% is the normal range on room air . A drop below 94% indicates hypoxemia and immediate assessment must be for airway and breathing.

IPD SHARING:
Plan to Share IPD: No